CLINICAL TRIAL: NCT07043829
Title: Effect of Consuming a Cimarrón Bean Extrudate Solution on Platelet Function and Postprandial Biochemical Parameters
Brief Title: Cimarrón Bean Extrudate Solution on Platelet Function and Biochemical Parameters
Acronym: CBE-SP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Talca (Other)
Collaborators: Centro de Estudios en Alimentos Procesados (Other)
Responsible Party: Principal Investigator, Iván Palomo González, Principal Investigator, University of Talca
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PCSAEPF29-2021
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Platelet Aggregation; Postprandial Glucose
Keywords: Phaseolus vulgaris; Platelet reactivity; Funtional food; Legume-base food; Platelet aggregation
MeSH Terms: interventions — Water

STUDY DESIGN:
Intervention Model Description: A single-group, open-label clinical trial in which all participants receive a single dose of a functional beverage containing 10 grams of Cimarrón bean extrudate dissolved in water. No placebo or comparator group is included. Outcomes are measured before and after the intervention within the same participants to assess acute changes in platelet function and postprandial glycemia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SAEP Intervention (Experimental): Participants will receive a single oral dose of 10 grams of Cimarrón bean extrudate dissolved in water. Platelet reactivity and postprandial glycemia will be measured before and after the intervention.
  Interventions: Dietary Supplement: SAEP (Solution of Cimarrón Bean Extrudate in Water)

INTERVENTIONS:
Dietary Supplement: SAEP (Solution of Cimarrón Bean Extrudate in Water) — A single oral dose of 10 grams of Cimarrón bean (Phaseolus vulgaris, variety Cimarrón) extrudate dissolved in 500 mL of water, consumed once under fasting conditions. Used to evaluate acute effects on platelet function and postprandial glycemia.

SUMMARY:
This non-randomized acute clinical trial evaluates the effect of consuming a water-based solution of Cimarrón bean extrudate on platelet function and postprandial glycemia in adults.

Participants will consume a single 10-gram dose of Cimarrón bean extrudate dissolved in water. Blood samples will be collected before and after the intervention to assess platelet reactivity using flow cytometry and to measure glucose levels through colorimetric spectrophotometry. The total intervention period will last approximately 8 hours. This study aims to explore whether the acute consumption of this legume-based functional product can influence hemostatic and glycemic responses in the postprandial state.

DETAILED DESCRIPTION:
This clinical trial aims to evaluate the acute effects of consuming a beverage made from Cimarrón bean extrudate on platelet function and postprandial blood glucose levels in adult participants. The study involves a single-arm, non-randomized, open-label design in which each participant will consume a single oral dose of 10 grams of Cimarrón bean extrudate dissolved in water (SAEP: Solution of Cimarrón Bean Extrudate in Water).

The trial includes baseline and post-intervention assessments of platelet reactivity using flow cytometry, employing specific agonists (CRP, TRAP, ADP) and labeled antibodies (anti-fibrinogen FITC, PE-CD61/CD62). Blood glucose levels will also be measured at multiple time points using colorimetric spectrophotometry to evaluate postprandial metabolic response.

The total study duration per participant is approximately 8 hours, including fasting baseline measurements, administration of the intervention, and postprandial monitoring. This study seeks to provide preliminary data on the potential hemostatic and glycemic effects of a legume-derived functional food ingredient in a controlled, acute setting.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participant
* Men and women aged 20-59 years
* Willingness to participate and provide written informend consent

Exclusion Criteria:

* Documented food allergies, especially ti legumes or beans
* Diagnosed liver, kidney, , autoinmune diseases or severe illnesses such as cancer.
* Diagnosed gastrointestinal diseases including inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis), celiac disease, or any condition causing chronic gastrointestinal symptoms such as malabsorption, persistent diarrhea, or gastrointestinal bleeding
* Use medication known to alter platelet funtion like, antiplatelet agents (aspirin, clopidogrel); Non-steroidal anti-inflamatory drugs (NSAID-Ibuprofen, naproxen); Anticoagulants (Warfarin, heparin, direct oral anticoagulant like rivaroxaban or apixaban); Selective serotonin reuptake inhibitors (SSRIs) and other drugs known to impact platelet aggregation or hemostasis.

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-03-13 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2025-06-19 (Actual)

PRIMARY OUTCOMES:
Change in platelet reactivity after acute consumption of SAEP | Baseline and 2 to 6 hours post-intervention
  Platelet reactivity will be assessed by flow cytometry using CRP, TRAP, and ADP as agonists, with fluorescent antibodies (anti-fibrinogen FITC and PE-CD61/CD62). Measurements will be performed before and after consumption of SAEP to evaluate acute changes in platelet activation.

SECONDARY OUTCOMES:
Change in postprandial blood glucose levels after consumption of SAEP | Baseline and up to 2 hours post-intervention
  Blood glucose concentrations will be measured at baseline and postprandial time, 2 hours after consuming 10 g of Cimarrón bean extrudate dissolved in water. The aim is to evaluate the glycemic response and potential glycemia-lowering effects of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan F Palomo Gonzalez, PhD. Biomedical Science, Principal Investigator — University of Talca; Eduardo J Fuentes Quinteros, PhD. Science research, Study Chair — University of Talca
Locations (1):
- Universidad de Talca, Talca, Maule Region, Chile

IPD SHARING:
Plan to Share IPD: Undecided
The plan to share individual participant data (IPD) has not yet been determined. The decision will depend on future publication plans, data management policies, and ethical considerations regarding participant privacy.